CLINICAL TRIAL: NCT05070546
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Safety and Immunogenicity of an Ad26.RSV.preF-based Vaccine in Adults Aged 18 to 59 Years, Including Those at High-risk for Severe RSV
Brief Title: A Study of an Ad26.RSV. preF-based Vaccine in Adults Aged 18 to 59 Years, Including Adults at High Risk for Severe RSV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109038; 2021-001909-77 (EudraCT Number); VAC18193RSV3006 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Infection Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort (C)1 Group (G)1: Healthy Adults, 18-59 Years (Respiratory Syncytial Virus [RSV] vaccine) (Experimental): Participants will receive a single intramuscular (IM) injection of study vaccine on Day 1.
  Interventions: Biological: Ad26.RSV.preF-based Vaccine
- C1 G2: Healthy Adults, 18-59 Years (Placebo) (Placebo Comparator): Participants will receive a single IM injection of matching placebo on Day 1.
  Interventions: Other: Placebo
- C2 G3: High Risk Adult, 18-59 Years (RSV Vaccine) (Experimental): Participants will receive a single IM injection of study vaccine on Day 1.
  Interventions: Biological: Ad26.RSV.preF-based Vaccine
- C2 G4: High Risk Adult, 18-59 Years (Placebo) (Placebo Comparator): Participants will receive a single IM injection of matching placebo on Day 1.
  Interventions: Other: Placebo
- C3 G5: Adults, 65 Years and Older (RSV Vaccine) (Experimental): Participants will receive a single IM injection of study vaccine on Day 1.
  Interventions: Biological: Ad26.RSV.preF-based Vaccine
- C3 G6: Adults, 65 Years and Older (Placebo) (Placebo Comparator): Participants will receive a single IM injection of matching placebo on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ad26.RSV.preF-based Vaccine — Participants will receive a single IM injection of an RSV vaccine.
  Arms: C2 G3: High Risk Adult, 18-59 Years (RSV Vaccine); C3 G5: Adults, 65 Years and Older (RSV Vaccine); Cohort (C)1 Group (G)1: Healthy Adults, 18-59 Years (Respiratory Syncytial Virus [RSV] vaccine)
Other: Placebo — Participants will receive a single IM injection of matching placebo.
  Arms: C1 G2: Healthy Adults, 18-59 Years (Placebo); C2 G4: High Risk Adult, 18-59 Years (Placebo); C3 G6: Adults, 65 Years and Older (Placebo)

SUMMARY:
The purpose of the study is to investigate the safety and immunogenicity of the Ad26.RSV.preF based vaccine in adults 18 to 59 years of age who are healthy or at risk for severe Respiratory Syncytial Virus (RSV) disease, compared to adults 65 years and above.

DETAILED DESCRIPTION:
RSV is an important cause of serious respiratory infections in adults aged 60 years and older, immunocompromised individuals, and those with underlying chronic cardiopulmonary conditions. The current study assess the safety and immunogenicity of the RSV vaccine in adults 18 to 59 years of age, including those who are at risk for severe RSV disease. The study comprises screening (pre-vaccination) and vaccination for each participant on Day 1, and a 6- month safety and immunogenicity follow-up period. The study duration will be up to 6 months per participant. Assessments like immunogenicity (such as humoral and cellular immune responses), safety (such as monitoring of AEs, physical examinations, and vital signs) and reactogenicity will be performed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be of a) non child bearing potential or b) of child bearing potential and practicing an acceptable and effective of contraception
* All participants of childbearing potential must: have a negative highly sensitive urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening; and have a negative highly sensitive urine beta-hCG pregnancy test immediately prior to each study vaccination (if screening and vaccination are not performed on the same day) Cohorts 1 and 2
* Participant is aged 18 to 59 years (inclusive) on the day of signing the informed consent form (ICF) and expected to be available for the duration of the study Cohort 2
* Has an existing chronic heart or lung condition, without hospitalizations or major medication class change (that is, new or stopped medications) within 30 days prior to screening, meeting the following criteria; a) cardiac disease: at least Class II symptoms per New York Heart Association classification or similar guidelines according to local practice, b) pulmonary disease: activity-restricting symptoms or use of long-term medications Cohort 3
* Participant is aged 65 years or older on the day of signing the ICF and expected to be available for the duration of the study
* Participant may have underlying illnesses such as hypertension, congestive heart failure, chronic obstructive pulmonary disease (COPD), type 2 diabetes, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are stable at the time of vaccination, and these conditions receive routine follow-up by the participant's healthcare provider

Exclusion Criteria:

* Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Abnormal function of immune system due to a clinical condition or treatment
* History of thrombosis with thrombocytopenia syndrome (TTS) or heparin-induced thrombocytopenia and thrombosis (HITT).
* Participant received or plans to receive: (a) licensed live attenuated vaccines - within 28 days before or after planned administration of study vaccine; and (b) other licensed (not live) vaccines - within 14 days before or after planned administration of study vaccine
* Received an respiratory syncytial virus (RSV) vaccine in a previous RSV vaccine study
* History of acute polyneuropathy (example, Guillain-Barre syndrome) or chronic idiopathic demyelinating polyneuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1124 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (23):
- United States (7):
  - Alliance for Multispeciality Research, Coral Gables, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Heartland Research Associates, an AMR Company, El Dorado, Kansas
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, New Orleans, Louisiana
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Tekton Research Inc., Yukon, Oklahoma
  - Alliance for Multispeciality Research, Knoxville, Tennessee
- Belgium (3):
  - Anima, Alken
  - C.H.U. St Pierre / Maladies Infectieuses, Brussels
  - Private Practice RESPISOM Namur, Namur
- Germany (7):
  - Emovis GmbH, Berlin
  - Klinische Forschung Berlin GbR, Berlin
  - Zentrum fuer klinische Forschung, Cologne
  - Klinische Forschung Dresden GmbH, Dresden
  - Clinical Research HamburggmbH, Hamburg
  - SIBAmed GmbH & Co. KG, Leipzig
  - Klinische Forschung Schwerin GmbH, Schwerin
- Spain (2):
  - Hosp Reina Sofia, Córdoba
  - Hosp Virgen de La Victoria, Málaga
- Sweden (4):
  - ProbarE i Lund AB, Lund
  - ClinSmart Sweden AB, Solna
  - ProbarE i Stockholm AB, Stockholm
  - Studieenheten Akademiskt Specialistcentrum Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] LaRoche JK, Lanier J, Alvarenga R, Collins M, Costelloe T, Chiau A, Whetherly H, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored in-human clinical trials: life cycle assessments of clinical trials spanning multiple phases and disease areas. BMJ Open. 2025 Feb 19;15(2):e085364. doi: 10.1136/bmjopen-2024-085364. PMID 39971605
- [Derived] Jastorff A, Gymnopoulou E, Salas J, Merrall E, Buntinx E, Martin C, Askling HH, Schenkenberger I, Yuste AC, Smith W, Sotolongo R, Von Engelhardt C, Bastian AR, Comeaux C, Ligtenberg N, Callendret B, Heijnen E. Safety and immunogenicity of the Ad26/protein preF RSV vaccine in adults aged 18 to 59 years with and without at-risk comorbidities for severe respiratory syncytial virus disease: A phase 3, randomized, controlled, immunobridging trial. Vaccine. 2025 Jan 1;43(Pt 1):126514. doi: 10.1016/j.vaccine.2024.126514. Epub 2024 Nov 12. PMID 39536455

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein: Healthy adult participants aged 18 to 59 years received a single intramuscular (IM) injection containing mixture of adenovirus serotype 26 respiratory syncytial virus pre-fusion conformation-stabilized F protein (Ad26.RSV.preF) 1*10^11 viral particles (vp) and RSV preF protein 150 micrograms (mcg) on Day 1.
- Group 2 (Cohort 1): Placebo: Healthy adult participants aged 18 to 59 years received a single IM injection of matching placebo on Day 1.
- Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein: High-risk adult participants aged 18 to 59 years received a single IM injection containing mixture of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg on Day 1.
- Group 4 (Cohort 2): Placebo: High-risk adult participants aged 18 to 59 years received a single IM injection of matching placebo on Day 1.
- Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein: Adult participants aged 65 years and older received a single IM injection containing mixture of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg on Day 1.
- Group 6 (Cohort 3): Placebo: Adult participants aged 65 years and older received a single IM injection of matching placebo on Day 1.
Period: Overall Study
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein | Group 6 (Cohort 3): Placebo
Started | 320 | 68 | 320 | 70 | 316 | 30
Vaccinated | 319 | 68 | 319 | 69 | 313 | 30
Completed | 310 | 65 | 309 | 68 | 308 | 29
Not Completed | 10 | 3 | 11 | 2 | 8 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 8 | 2 | 7 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Randomized but not vaccinated | 1 | 0 | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received study vaccine, regardless of the occurrence of protocol deviations and vaccine type (study vaccine or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein | Group 6 (Cohort 3): Placebo | Total
Number analyzed (Participants) | 319 | 68 | 319 | 69 | 313 | 30 | 1118
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.33) | 38.4 (12.34) | 44.4 (11.81) | 44.6 (11.58) | 71.1 (4.74) | 71.2 (5.1) | 50.6 (17.27)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 319 | 68 | 319 | 69 | 0 | 0 | 775
  From 65 and over | 0 | 0 | 0 | 0 | 313 | 30 | 343
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 40 | 174 | 39 | 181 | 21 | 648
  Male | 126 | 28 | 145 | 30 | 132 | 9 | 470
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 10 | 40 | 9 | 19 | 2 | 122
  Not Hispanic or Latino | 274 | 57 | 276 | 60 | 289 | 28 | 984
  Unknown or Not Reported | 3 | 1 | 3 | 0 | 5 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 2 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Black or African American | 24 | 4 | 7 | 1 | 9 | 0 | 45
  White | 289 | 64 | 308 | 68 | 303 | 29 | 1061
  More than one race | 4 | 0 | 0 | 0 | 0 | 1 | 5
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 178 | 36 | 38 | 5 | 18 | 3 | 278
  GERMANY | 0 | 0 | 175 | 38 | 88 | 11 | 312
  SPAIN | 0 | 0 | 15 | 5 | 0 | 0 | 20
  SWEDEN | 33 | 8 | 50 | 15 | 160 | 11 | 277
  UNITED STATES | 108 | 24 | 41 | 6 | 47 | 5 | 231

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 2: Number of Participants With Solicited Local Adverse Events (AEs)
Description: Number of participants with solicited local AEs at 7 days post-vaccination in Cohorts 1 and 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were predefined local events (at the injection site: erythema, pain/tenderness and swelling) that were by definition considered as related to the study vaccine and collected within 7 days after vaccination.
Time Frame: 7 days after vaccination on Day 1 (Day 8)
Population: Full analysis set (FAS) included all participants who received study vaccine, regardless of the occurrence of protocol deviations and vaccine type (study vaccine or placebo). Here 'N' (number of participants analysed) signifies number of participants who were evaluable for this outcome measure. This outcome measure was planned to be analysed for specified cohorts only.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo
Number analyzed (Participants) | 316 | 68 | 318 | 68
Participants | 273 | 10 | 276 | 15

2. Primary Outcome: Cohorts 1 and 2: Number of Participants With Solicited Systemic AEs
Description: Number of participants with solicited systemic AEs at 7 days post-vaccination in Cohorts 1 and 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited systemic AEs including pyrexia, headache, fatigue, myalgia and nausea were collected within 7 days after vaccination.
Time Frame: 7 days after vaccination on Day 1 (Day 8)
Population: FAS included all participants who received study vaccine, regardless of the occurrence of protocol deviations and vaccine type (study vaccine or placebo). Here 'N' (number of participants analysed) signifies number of participants who were evaluable for this outcome measure. This outcome measure was planned to be analysed for specified cohorts only.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo
Number analyzed (Participants) | 316 | 68 | 318 | 68
Participants | 277 | 33 | 275 | 40

3. Primary Outcome: Cohorts 1 and 2: Number of Participants With Unsolicited AEs
Description: Number of participants with unsolicited AEs post-vaccination in Cohorts 1 and 2 were reported. An AE was defined as any untoward medical occurrence in a participant participating in a clinical study that did not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were defined as all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: 28 days after vaccination on Day 1 (Day 29)
Population: FAS included all participants who received study vaccine, regardless of the occurrence of protocol deviations and vaccine type (study vaccine or placebo). This outcome measure was planned to be analysed for specified cohorts only.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo
Number analyzed (Participants) | 319 | 68 | 319 | 69
Participants | 111 | 13 | 85 | 12

4. Primary Outcome: Cohorts 1, 2, and 3: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with SAEs post-vaccination were reported. An AE was defined as any untoward medical event that occurred in a participant administered an investigational product, and it did not necessarily indicated only events with clear causal relationship with the relevant investigational product. SAE was defined as any AE that resulted in: death, persistent or significant disability/incapacity, required inpatient hospitalization or prolongation of existing hospitalization, was life-threatening experience, was a congenital anomaly/birth defect and would jeopardize participant and/or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: 6 months after vaccination on Day 1 (Day 183)
Population: FAS included all participants who received study vaccine, regardless of the occurrence of protocol deviations and vaccine type (study vaccine or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein | Group 6 (Cohort 3): Placebo
Number analyzed (Participants) | 319 | 68 | 319 | 69 | 313 | 30
Participants | 1 | 1 | 10 | 0 | 13 | 1

5. Primary Outcome: Cohorts 1, 2, and 3: Number of Participants With Adverse Events of Special Interest (AESI)
Description: Number of participants with AESI post-vaccination were reported. AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with thrombocytopenia syndrome (TTS) was considered as an AESI.
Time Frame: 6 months after vaccination on Day 1 (Day 183)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein | Group 6 (Cohort 3): Placebo
Number analyzed (Participants) | 319 | 68 | 319 | 69 | 313 | 30
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Cohorts 1 (Group 1), 2 (Group 3), and 3 (Group 5): Respiratory Syncytial Virus (RSV) A2 Strain Neutralizing Antibody Titers
Description: RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay and were expressed as 50% inhibitory concentration (IC50) units.
Time Frame: 14 days after vaccination on Day 1 (Day 15)
Population: The Per-protocol Immunogenicity (PPI) set included all randomised participants on Day 15 who received study vaccine and for whom immunogenicity data were available. Here 'N' (number of participants analysed) signifies number of participants who were evaluable for this outcome measure. This outcome measure was planned to be analysed for specified arms only. As planned, combined data of participants aged 18-59 years Cohorts 1 (Group 1) and 2 (Group 3) has been reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Group 1 (Cohort 1) and Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein: Healthy (Group 1) and high-risk adult (Group 3) participants aged 18 to 59 years received intramuscular (IM) injection containing mixture of adenovirus serotype 26 pre-fusion conformation-stabilized F protein (Ad26.RSV.preF) 1*10^11 viral particles (vp) and respiratory syncytial virus prefusion F-protein (RSV preF protein) 150 micrograms (mcg) on Day 1.
Arm/Group | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein | Group 1 (Cohort 1) and Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein
Number analyzed (Participants) | 301 | 290 | 602
Titers | 7095 [6261 to 8042] | 4596 [4059 to 5204] | 6491 [5847 to 7206]
Statistical Analysis 1: Comparison: Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein vs Group 1 (Cohort 1) and Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein; Test type: Non-Inferiority — Non-inferiority of Cohort 3 (Group 5) versus Cohorts 1 (Group 1) and 2 (Group 3) in terms of RSV A2 Strain neutralizing antibody titers against 14 days after vaccination, using a non-inferiority margin of 0.67 for the GMT ratio (Cohort 3 [Group 5]/Cohort 1[Group1] and 2 [Group 3]); Geometric Mean Ratio; Geometric Mean Ratio = 1.41, 95% CI 2-sided [1.25 to 1.60]
Statistical Analysis 2: Comparison: Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein vs Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein; Test type: Non-Inferiority — Non-inferiority of Cohort 3 (Group 5) versus Cohort 2 (Group 3 in terms of RSV A2 Strain neutralizing antibody titers against 14 days after vaccination, using a non-inferiority margin of 0.67 for the GMT ratio (Cohort 3 [Group 5]/Cohort 2 [Group 3]); Geometric Mean Ratio; Geometric mean ratio = 1.54, 95% CI 2-sided [1.34 to 1.78]

7. Primary Outcome: Cohorts 1 (Group 1), 2 (Group 3), and 3 (Group 5): Percentage of Participants With Seroresponse as Assessed by Virus Neutralizing Assay (VNA-A2)
Description: Percentage of participants with seroresponse as assessed by VNA-A2 strain were reported. Seroresponse was defined as a 4-fold increase from baseline in Day 15 VNA A2 antibody titers.
Time Frame: 14 days after vaccination on Day 1 (Day 15)
Population: PPI set included all randomized participants who received study vaccine and for whom immunogenicity data were available. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. This outcome measure was planned to be analysed for specified arms only. As planned, combined data of participants aged 18-59 years Cohorts 1 (Group 1) and 2 (Group 3) has been reported.
Measure: Number; unit: percentage of participants
Groups:
- Cohorts 1(Group 1) and 2 (Group 3): Ad26.RSV.preF and RSV preF Protein: Healthy (Group 1) and high-risk adult (Group 3) participants aged 18 to 59 years received intramuscular (IM) injection containing mixture of adenovirus serotype 26 pre-fusion conformation-stabilized F protein (Ad26.RSV.preF) 1*10^11 viral particles (vp) and respiratory syncytial virus prefusion F-protein (RSV preF protein) 150 micrograms (mcg) on Day 1.
Arm/Group | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein | Cohorts 1(Group 1) and 2 (Group 3): Ad26.RSV.preF and RSV preF Protein
Number analyzed (Participants) | 300 | 290 | 602
percentage of participants | 88 | 82.41 | 89.37
Statistical Analysis 1: Comparison: Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein vs Cohorts 1(Group 1) and 2 (Group 3): Ad26.RSV.preF and RSV preF Protein; Test type: Non-Inferiority — Non-inferiority of Cohort 3 (Group 5) versus Cohorts 1 (Group 1) and 2 (Group 3) in terms of RSV A2 Strain neutralizing antibody titers against 14 days after vaccination, using a non-inferiority margin of -10% for the GMT ratio (Cohort 3 [Group 5]/Cohort 1[Group1] and 2 [Group 3]); Difference in Seroresponse rate; Difference in Seroresponse rate = 5.4, 95% CI 2-sided [0.3 to 10.9]
Statistical Analysis 2: Comparison: Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein vs Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein; Test type: Non-Inferiority — Non-inferiority of Cohort 3 (Group 5) versus Cohorts 1 (Group 1) and 2 (Group 3) in terms of RSV A2 Strain neutralizing antibody titers against 14 days after vaccination, using a non-inferiority margin of -10% for the GMT ratio (Cohort 3 [Group 5]/Cohort 2 [Group 3]); Difference in Seroresponse rate; Difference in Seroresponse rate = 4.4, 95% CI 2-sided [-1.6 to 10.5]

8. Secondary Outcome: Cohorts 1, 2, and 3: Geomteric Mean Titers (GMTs) of RSV Fusion Protein (F-protein) Antibodies as Assessed by Enzyme-linked Immunosorbent Assay (ELISA)- Pre-Fusion
Description: GMTs of RSV Fusion Protein (PreF) antibodies as assessed by ELISA-Pre-Fusion at Day 15 were reported.
Time Frame: 14 days after vaccination on Day 1 (Day 15)
Population: PPI set included all randomised participants who received study vaccine and for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per liter (EU/L)
Groups:
- Cohort 3: Adults: RSV Vx (Group 5): Adult participants aged 65 years and older received IM injection containing Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg on Day 1 of vaccination.
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo | Cohort 3: Adults: RSV Vx (Group 5) | Group 6 (Cohort 3): Placebo
Number analyzed (Participants) | 302 | 64 | 301 | 61 | 290 | 29
ELISA units per liter (EU/L) | 4662 [4350 to 4997] | 246 [214 to 284] | 5175 [4808 to 5569] | 283 [246 to 326] | 3864 [3559 to 4196] | 240 [203 to 285]

ADVERSE EVENTS:
Time Frame: Up to Day 183
Description: Full analysis set included all participants who received study vaccine, regardless of the occurrence of protocol deviations and vaccine type (study vaccine or placebo).
Arm/Group | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein | Group 2 (Cohort 1): Placebo | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein | Group 4 (Cohort 2): Placebo | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein | Group 6 (Cohort 3): Placebo
All-Cause Mortality (participants affected / at risk) | 0/319 | 0/68 | 0/319 | 0/69 | 0/313 | 1/30
Serious Adverse Events (participants affected / at risk) | 1/319 | 1/68 | 10/319 | 0/69 | 13/313 | 1/30
Other Adverse Events (participants affected / at risk) | 77/319 | 5/68 | 50/319 | 8/69 | 32/313 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein (N=319) | Group 2 (Cohort 1): Placebo (N=68) | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein (N=319) | Group 4 (Cohort 2): Placebo (N=69) | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein (N=313) | Group 6 (Cohort 3): Placebo (N=30)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhagic Fever with Renal Syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Meningitis Aseptic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bladder Cancer Stage 0, with Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Her2 Positive Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Facial Paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Testicular Torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Cohort 1): Ad26.RSV.preF and RSV preF Protein (N=319) | Group 2 (Cohort 1): Placebo (N=68) | Group 3 (Cohort 2): Ad26.RSV.preF and RSV preF Protein (N=319) | Group 4 (Cohort 2): Placebo (N=69) | Group 5 (Cohort 3): Ad26.RSV.preF and RSV preF Protein (N=313) | Group 6 (Cohort 3): Placebo (N=30)
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 8 | 0 | 2 | 0 | 2 | 0
Chills (General disorders) | 60 | 1 | 31 | 1 | 15 | 0
Covid-19 (Infections and infestations) | 8 | 1 | 4 | 3 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 9 | 3 | 9 | 1
Sinusitis (Infections and infestations) | 7 | 0 | 1 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 1 | 3 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 4 | 2 | 0 | 2 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 8 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT05070546/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT05070546/SAP_001.pdf